CLINICAL TRIAL: NCT02170168
Title: The Orkdal Model. Development, Implementation and Evaluation of Collaboration Between Specialist and Community Care Within Palliative Cancer Care
Brief Title: The Orkdal Model. Collaboration Between Specialist and Community Care Within Palliative Cancer Care
Status: Completed | Type: Observational
Sponsor: St. Olavs Hospital (Other)
Collaborators: The Coordination Unit in the Orkdal region (SIO) (Unknown); Helse Møre og Romsdal HF (Other Government); Norwegian University of Science and Technology (Other)
Responsible Party: Sponsor
Other Study IDs: 2014/212
Record Dates: First submitted 2014-06-19; First posted 2014-06-23 (Estimated); Last update posted 2023-04-13 (Actual); Status verified 2023-04

CONDITIONS: Neoplasms
Keywords: Community health services; Models, organizational; Referral and consultation; Palliative medicine; Terminal care
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (6):
- Orkdal region patients: cancer patients participating in a integrated palliative care program for diagnostics, treatment, care and follow-up in and between hospital care and 13 municipalities
  Interventions: Other: integrated palliative care program
- Romsdal county patients: control palliative care cancer patients in standard care, i.e. a local hospital in the county of Møre and Romsdal, Molde Hospital, and nine districts
- Orkdal region carers: carers of cancer patients participating in a integrated palliative care program for diagnostics, treatment, care and follow-up in and between hospital care and 13 municipalities
  Interventions: Other: integrated palliative care program
- Romsdal county carers: carers of cancer patients receiving standard care, i.e. in a local hospital in the county of Møre and Romsdal, Molde Hospital, and community care in nine districts
- Orkdal region health care providers: Health care providers for cancer patients participating in a integrated palliative care program for diagnostics, treatment, care and follow-up in and between hospital care and 13 municipalities
  Interventions: Other: integrated palliative care program
- Romsdal county health care providers: Health care providers for cancer patients receiving standard care, i.e. in a local hospital in the county of Møre and Romsdal, Molde Hospital, and community care in nine districts

INTERVENTIONS:
Other: integrated palliative care program — a standardised care pathway, an educational programme and information to general public, patients and their carers
  Groups: Orkdal region carers; Orkdal region health care providers; Orkdal region patients

SUMMARY:
The overall aim of this project is to deliver better health care services through improved coordination of cancer care within specialist care (at the local hospital Orkdal Hospital) and community care (13 municipalities in the Orkdal region, Norway), and between these two levels in the health care system. "The Orkdal model" is developed and will be implemented and evaluated within cancer care. Cancer patients living in one of the 12 municipalities participating in the formal collaboration "Samhandlingsenheten i Orkdalsregionen" (SIO), or the municipality of Oppdal, having metastatic and/or loco-regional disease will be included in the study. Carers and health care providers will be included as well. Results from this project will be transferable to other parts of Norway and/or to other countries as well as to patients with other diagnoses causing complex conditions, such as chronic heart-, lung- and neurological disease.

DETAILED DESCRIPTION:
This study will be a prospective controlled observational pre-post study. The intervention consists of three parts: a standardised care pathway, an educational programme and information to general public, patients and their carers. Data from patients, carers and health care providers (physicians, nurses and nurse assistants) will be collected before the model is implemented (pre-intervention part) and after final implementation (post-intervention part). In addition, a comparison with a similar patient population, carers and health care providers will be conducted. A local hospital in the county of Romsdal and community care in the same region will be used as control.

Added January 2020: The study was in 2018 extended to also evaluate the effect of implementing "advance care planning" in the county of Møre and Romsdal. Møre and Romsdal started implementation of "advance care planning" in January 2018. The evaluation of "advance care planning in Møre and Romsdal" has the same endpoints as the evaluation of the Orkdal model trial.

Added December 17th, 2021: Inclusion of participants (patients, carers and healthcare professionals) is from Sept 2018 to March 2021. Follow-up ends in Sept. 2022.

ELIGIBILITY:
Inclusion Criteria (Patients):

* Advanced loco-regional disease and/or metastatic cancer disease
* For the intervention group in the Orkdal region: Inhabitant of one of the following thirteen districts: Surnadal, Halsa, Rindal, Hemne, Orkdal, Frøya, Hitra, Snillfjord, Agdenes, Meldal, Rennebu, Skaun, and Oppdal
* For the intervention group in the Romsdal region: Inhabitiant of one of the following nine districts: Aukra, Molde, Eide, Vestnes, Sunndal, Fræna, Midsund, Nesset, Rauma
* Acceptance of participation, based on information about the study and that participation is voluntary. Documented by a signed consent form.
* Able to comply with the study procedures
* Able to read and write Norwegian

Inclusion criteria (Carers) (a carer a person identified as such by the patient)

* the patient is eligible for the study
* the patient has given his or her consent to allow the study nurse to approach the carer to participate in the study
* the patient has identified the carer to be approached
* acceptance of participation, based on information about the study and that participation is voluntary. Documented by a signed consent form.

Inclusion Criteria (Health care providers)

* has accepted to participate in the study
* Acceptance of participation, based on information about the study and that participation is voluntary. Documented by an electronically signed consent form.

Exclusion Criteria (Patients):

* Receiving anti-cancer treatment with curative intent

Exclusion Criteria (Carers)

* not able to complete the assessments

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Cancer patients in need of palliative care, inhabitants of one of 22 municipalities in Central Norway, carers (1 per patient) and health care providers (community care and 2 regional hospitals)
Sampling Method: Non-Probability Sample
Enrollment: 969 (Actual)
Dates: Start 2014-11 (Actual); Primary Completion 2022-03-31 (Actual); Study Completion 2022-09-30 (Actual)

PRIMARY OUTCOMES:
proportion of patient's time spent at home the last 3 months of life | 3 years
  time in days
carers' health related quality of life (HRQOL) 6 months after patient's death | 3 years
  as measured by the total score of the RAND-Short Form-36

SECONDARY OUTCOMES:
Number of home deaths | 3 years
Use of tumor directed treatment the last 3 months of life | 3 years
  radiotherapy and chemotherapy
change over time in health care providers' knowledge and skills | 3 years

OTHER OUTCOMES:
Patient reported health-related quality of life | 3 years
  measured by the total score of the European Organisation for the Research and Treatment of Cancer Core Quality of Life Questionnaire EORTC QLQ C15
place of death | 3 years
  if place of death is in accordance with patients' wish as reported at inclusion
distribution of health care services usage | 3 yeart
  between specialist and community care
total cost per patient | 3 years
share of specialist and community care costs | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Jo-Åsmund Lund, MD PhD, Study Director — St. Olavs Hospital
Locations (25):
- Norway (25):
  - Agdenes community care, Agdenes
  - Aukra community care, Aukra
  - Eide community care, Eide
  - Fræna community care, Fræna
  - Frøya community care, Frøya
  - Halsa community care, Halsa
  - Hemne community care, Hemne
  - Hitra community care, Hitra
  - Meldal community care, Meldal
  - Midsund community care, Midsund
  - Molde community care, Molde
  - Molde Hospital, Molde
  - Nesset community care, Nesset
  - Oppdal community care, Oppdal
  - Oppdal community care, Orkdal
  - Orkdal Hospital, Orkdal
  - Rauma community care, Rauma
  - Rennebu community care, Rennebu
  - Rindal community care, Rindal
  - Skaun community care, Skaun
  - Snillfjord community care, Snillfjord
  - Sunndal community care, Sunndal
  - Surnadal community care, Surnadal
  - St Olavs Hospital, Trondheim
  - Vestnes community care, Vestnes

REFERENCES:
- [Derived] Brenne AT, Lohre ET, Knudsen AK, Lund JA, Thronaes M, Driller B, Brunelli C, Kaasa S. Standardizing Integrated Oncology and Palliative Care Across Service Levels: Challenges in Demonstrating Effects in a Prospective Controlled Intervention Trial. Oncol Ther. 2024 Jun;12(2):345-362. doi: 10.1007/s40487-024-00278-3. Epub 2024 May 14. PMID 38744750
- [Derived] Driller B, Talseth-Palmer B, Hole T, Stromskag KE, Brenne AT. Cancer patients have a reduced likelihood of dying in hospital with advance care planning in primary health care and a summarizing palliative plan: a prospective controlled non-randomized intervention trial. Scand J Prim Health Care. 2024 Sep;42(3):471-482. doi: 10.1080/02813432.2024.2346131. Epub 2024 Apr 25. PMID 38662520